CLINICAL TRIAL: NCT00805623
Title: Partial Blinded Controlled Study to Compare SucroseVs Water, With and Without Pacifier as Pain Reliever During Venous Puncture in Infants 3-12 Months Old
Brief Title: Sucking and Sucrose as Pain Relief for Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Schneider Children's Medical Center of Israel, Schneider Children's Medical Center of Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 004994
Record Dates: First submitted 2008-12-07; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Pain
Keywords: sucrose; sucking; pain relief; infant; require venous puncture
MeSH Terms: conditions — Pain | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AW (No Intervention): no pacifier , no sucrose
- AS (Active Comparator): sucrose without pacifier
  Interventions: Dietary Supplement: sucrose
- PW (No Intervention)
- PS (Experimental): Pacifier and sucrose interventional
  Interventions: Dietary Supplement: sucrose

INTERVENTIONS:
Dietary Supplement: sucrose — 1 cc of sucrose 33.5% with or without pacifier
  Other Names: no other name
  Arms: AS; PS

SUMMARY:
Sucking and sucrose have been shown to reduce pain during venous puncture in neonates. Our study is designed to see if sucking and sucrose relieve pain during venous puncture in infants age 3-12 months.

DETAILED DESCRIPTION:
100 infants age 3-12 months old without neurologic, developmental or cardio-respiratory impairment, needing venous puncture for IV access, or blood aspiration, will be randomly assigned to one of 2 groups - with or without pacifier. During the puncture, each patient with pacifier will receive either 1 cc of water or 1 cc of sucrose (the solutions prepared and marked blindly) . Each patient without pacifier 2 will receive 1 cc of water without pacifier,will receive either 1 cc of water or 1 cc of sucrose (the solutions prepared and marked blindly). FLACC pain score will be used for apin assessment before, during and after the puncture.Comparison of the four groups will be done after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* age 3-12 months
* hospitalized in pediatric ward B
* need venous puncture

Exclusion Criteria:

* neurological deficit
* developmental delay
* Cyanotic heart disease
* symptomatic respiratory disease
* known problematic venous access

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-08 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
reduced pain scoring | 10 minutes

SECONDARY OUTCOMES:
better Parent's scoring to the child's behavior | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Efrat, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel